CLINICAL TRIAL: NCT06577818
Title: Sustained Inflation and Chest Compression Versus 3:1 Chest Compression to Ventilation Ratio During Cardiopulmonary Resuscitation of Asphyxiated Newborns - a Multi-centre, International Cluster Randomized Control Trial
Brief Title: Sustained Inflation and Chest Compression vs 3:1 C:V Ratio in Asphyxiated Newborns
Acronym: SUR1VE-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00145624
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CC+SI (Chest compression during sustained inflation) (Experimental): CC+SI Group (Intervention group): Newborns randomized to "CC+SI" will receive CPR with a SI using a peak inflation pressure (PIP) of 30cmH2O while receiving CC. The PIP was chosen based on our animal studies and two previous clinical trials. CC will be performed at a rate of minimum 90/min. Each SI will be delivered for duration of 30sec with a 1 sec pause between the next SI for 30sec is started while CCs are continued. After 2x30sec CC+SI (total of 60sec), Heart rate (HR) will be assessed: A HR <60/min means CC+SI is continued for another 60sec (2x30sec CC+SI), followed by another HR assessment. If HR >60/min, CC are stopped (current standard of care). CC+SI will continued until ROSC.
  Interventions: Procedure: CC+SI (Chest compression during sustained inflation)
- 3:1 C:V (3:1 Compression:Ventilation ratio) (Active Comparator): 3:1 C:V Group (Control group - Standard of Care): Newborns randomized to "3:1 C:V" will receive a CC rate of 90/min and 30 ventilations/min as per current resuscitation guidelines. The PIP used for the 30 inflations will also be 30cmH2O) as per current resuscitation guidelines. Every 60sec, a HR assessment as per neonatal guidelines will be performed to assess if HR is <60/min - continue CC or >60/min - stop CC (current standard of care). 3:1 C:V will be continued until ROSC.
  Interventions: Procedure: 3:1 C:V (3:1 Compression:Ventilation ratio)

INTERVENTIONS:
Procedure: CC+SI (Chest compression during sustained inflation) — CC+SI (Chest compression during sustained inflation)
  Arms: CC+SI (Chest compression during sustained inflation)
Procedure: 3:1 C:V (3:1 Compression:Ventilation ratio) — 3:1 C:V Group (Control group - Standard of Care): Newborns randomized to "3:1 C:V" will receive a CC rate of 90/min and 30 ventilations/min as per current resuscitation guidelines. The PIP used for the 30 inflations will also be 30cmH2O) as per current resuscitation guidelines. Every 60sec, a HR assessment as per neonatal guidelines will be performed to assess if HR is <60/min - continue CC or >60/min - stop CC (current standard of care). 3:1 C:V will be continued until ROSC.
  Arms: 3:1 C:V (3:1 Compression:Ventilation ratio)

SUMMARY:
Newborn infants who require cardiopulmonary resuscitation at birth receive chest compression using a 3-Compression to 1-Ventilation (3:1 C:V) ratio. However, the optimal chest compression technique during cardiopulmonary resuscitation is uncertain and identified as a critical gap in evidence.

The International Consensus Statement advises to use the 3:1 C:V ratio based on animal studies, and states that there are no clinical trials to support this approach and called for more research. There continues to be uncertainty about the optimal chest compression technique during cardiopulmonary resuscitation.

This trial will compare if in newborn infants with cardiac arrest in the delivery room does providing CC+SI (a new chest compression technique) compared to 3:1 C:V decreases the incidence of all mortality within the initial hospital stay.

This will be a multi-centre international cluster randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Newborns with gestational age born between 28 to 43 weeks based on best available obstetrical estimate
* Newborns designated to receive full resuscitation, i.e., parental request or pre-determined decision to provide only comfort care at birth
* No known major congenital or chromosomal malformation. All newborns who meet inclusion criteria will be enrolled as the centres agreed to change their local hospital policy during the trial. The inclusion criteria are designed to be pragmatic and provide useful knowledge translation for most of the patient population in the future.

Exclusion Criteria:

- Newborns born outside of study centers and transported to centers after delivery.

Sex, race, and ethnicity are not part of the exclusion criteria for this trial, and as such it should represent the combined demographics of all centers involved.

Max Age: 40 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 554 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2031-07-01 (Estimated); Study Completion 2033-07-01 (Estimated)

PRIMARY OUTCOMES:
Neonatal mortality | 0-40 days after birth
  All mortality within the initial hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schmolzer, Principal Investigator — University of Alberta
Locations (1):
- Royal Alexandra Hospital, Edmonton, Canada

IPD SHARING:
Plan to Share IPD: Undecided